CLINICAL TRIAL: NCT04395196
Title: A Randomized, Double-Blind, Placebo-controlled Clinical Trial of Choline Supplementation During Pregnancy to Mitigate Adverse Effects of Prenatal Alcohol Exposure on Growth and Cognitive Development
Brief Title: RCT of Prenatal Choline Supplementation During Pregnancy to Mitigate Adverse Effects of Prenatal Alcohol Exposure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of Cape Town (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Sandra W. Jacobson, Ph.D, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AA028053 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Fetal Alcohol Spectrum Disorders; Fetal Alcohol Syndrome
Keywords: Prenatal Alcohol Exposure; Choline Supplementation; Infant Neurodevelopment; Growth
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose choline supplementation (Active Comparator): 2 g choline cation
  Interventions: Dietary Supplement: Choline bitartrate
- Placebo (Placebo Comparator): Placebo identical to active treatment in appearance, taste, and smell.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Choline bitartrate — Provided in beverage form
  Arms: High-dose choline supplementation
Dietary Supplement: Placebo — Provided in beverage form
  Arms: Placebo

SUMMARY:
Although the adverse effects associated with prenatal alcohol exposure (PAE) are well known, many women continue to drink heavily during pregnancy, putting their infants at risk for fetal alcohol spectrum disorders. Animal studies have shown that choline supplementation can mitigate effects of PAE on growth and development. Choline, an essential nutrient, serves as a methyl-group donor for DNA methylation and is a constituent of the neurotransmitter acetylcholine and a precursor to major components of cell membranes. In an R21 feasibility trial, 70 heavy drinkers were randomly assigned to receive a daily dose of 2g of choline or a placebo from initiation of antenatal care to delivery in Cape Town, South Africa, where the incidence of heavy drinking during pregnancy and fetal alcohol syndrome are among the highest in the world. When compared with infants in the placebo arm, infants in the choline-treated arm were more likely to meet criterion for eyeblink conditioning, demonstrated markedly better recognition memory on the Fagan Test of Infant Intelligence, which is known to have predictive validity for school-age IQ, and had better postnatal gains in weight and head circumference. Key features of this study included the higher choline dose (4.4 times adequate intake (AI), compared to 1.7-2.5 in previous human studies) and initiation of treatment early in pregnancy. We are now conducting a fully-powered, double-blind, randomized, placebo-controlled choline supplementation trial in heavy drinking pregnant women from a rural community in South Africa (1) to assess the effectiveness of maternal choline supplementation during pregnancy to mitigate effects of PAE on three primary outcomes: infant recognition memory and postnatal growth restriction (weight and head circumference); (2) to assess the efficacy of this supplementation for mitigating alcohol effects on the following secondary outcomes: infant eyeblink conditioning, postnatal length, and information processing speed; (3) to use innovative methods in causal inference analysis to examine protocol adherence as an important source of variation in treatment efficacy and to identify sociodemographic factors associated with non-compliance in order to facilitate implementation of the intervention protocol in clinical settings; and (4) in exploratory analyses, to examine whether maternal choline supplementation is particularly effective in women with lower dietary choline intake or poor nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 yr
* ≤20 wk gestation
* Singleton pregnancy
* Currently heavy drinking (average of ≥15 ml AA/day or binge drinking (≥4 standard drinks/occasion) on at least 1.5 occasions/month on average since becoming pregnant)
* Current choline dietary intake <1 g/day
* Language fluency in English or Afrikaans

Exclusion Criteria:

* Use of methamphetamine or other illicit drugs other than marijuana during the past year
* HIV positive
* Pharmacologic treatment for a serious pre-existing medical condition (e.g., diabetes, hypertension, epilepsy, or cardiac problems)
* Having another child enrolled in the trial from a previous pregnancy
* Plans for mother or child to move away from the area prior to study completion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Infant recognition memory | 12 months
  Novelty preference from the Fagan Test of Infant Intelligence
Postnatal infant weight gain | 6.5 months
Postnatal growth in infant head circumference | 6.5 months

SECONDARY OUTCOMES:
Infant information processing speed | 12 months
  Processing speed on the Fagan Test of Infant Intelligence
Postnatal growth in infant length | 6.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra W Jacobson, PhD, Principal Investigator — Wayne State University; Joseph L Jacobson, PhD, Principal Investigator — Wayne State University; Ernesta M Meintjes, PhD, Principal Investigator — University of Cape Town Faculty of Health Sciences; R. Colin Carter, MD, MMSc, Principal Investigator — Columbia University Vagelos College of Physicians and Surgeons
Locations (1):
- University of Cape Town Faculty of Health Sciences, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
We will make data collected in this study publicly available in accordance with the policies laid out in the NIH/National Institute on Alcohol Abuse and Alcoholism (NIAAA) Data-Sharing Policy for Human Subjects Grants Research Funded by the NIAAA (NOT-AA-18-010; https://grants.nih.gov/grants/guide/notice-files/NOT-AA-18- 010.html). Individual participant data relating to the chief aims of this study data obtained with NIAAA funding will be uploaded to the NIAAA Data Archive (NIAAADA). Only de-identified data will be available to the NIAAADA. A data dictionary will also be available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Per NIAAA policies, data will be made available for sharing with researchers 2 years after the end of the grant or 2 years after the end date of a no-cost-extension, if issued. The end date for data requests will be determined by NIAAA policies.
Access Criteria: Per NIAAA guidelines, for research purposes, "investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NIAAADA data by submitting a data access request in accordance with applicable NIAAADA policies (see https://ndar.nih.gov/access.html for sample policies). Data requests will be reviewed and granted by an NIAAA Data Access Committee." The study protocol, statistical analysis plan, and analytic code may be shared by requests to PI Sandra W. Jacobson, PhD.